CLINICAL TRIAL: NCT02954614
Title: Active Play -an After-school-program Intervention to Promote Physical Activity and Health-related Quality of Life in Young Children
Brief Title: Active Play in After School Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Principal Investigator, Kirsti Riiser, Phd, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 46008
Record Dates: First submitted 2016-10-26; First posted 2016-11-03 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Physical Activity; Activity Play; Motor Activity; Quality of Life; Autonomy; Competence; Children; After-School Program
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Active play in after school programs (ASP). Training program for ASP staff.
  Interventions: Behavioral: Active play in after school programs (ASP)
- Control group (No Intervention): ASP as usual.

INTERVENTIONS:
Behavioral: Active play in after school programs (ASP) — * A 15 hour training-program for ASP-staff aimed to increase active play and physical activity among children in ASPs. The program includes lectures, guided discussions and practical tasks focusing on increasing the staffs competence in how to support active play and PA among all children in the ASP
  * A 8 hour course for local physiotherapists enabling them to guide ASP-staff during parts of the intervention period
  Arms: Intervention group

SUMMARY:
Background: Physical activity (PA) is a key component in health promotion and prevention of overweight. Interventions delivered in after-school programs (ASP) have the potential to become a means of ensuring PA among young schoolchildren. This requires a motivational climate, allowing for self-determination and the intrinsic values of the activity, on the activity's character of play. ASP staff could be trained in stimulating all children in physical activities in their everyday life. Physiotherapists in primary care possess knowledge of motor development and learning, and are important contributors to an ASP-based physical activity intervention.

Aim: To develop a complex intervention that emphasizes physical activity play, and to examine through a cluster-randomized trial the extent to which the intervention promotes PA and health-related quality of life and prevents overweight in a population of young children. We aim to increase the knowledge and autonomy supportive skills among ASP staff members, enabling them to promote physical activity through play among all first graders in ASP.

In addition to investigate if the children benefit from receiving autonomy support, we aim to study whether the ASP staff themselves benefit from giving autonomy support in terms of increased need satisfaction and autonomous motivation for work.

The intervention: Includes training of ASP-staff members in the fundamental principles of self-determination theory and practical applications for motivating young children in PA through play. Information will be given on the benefits of a physically active lifestyle and the staff will be encouraged to map opportunities for PA in their local ASP and to incorporate strategies to increase PA through play among the children throughout the day.

Methods/design: A complex intervention using a mixed methods approach will be developed and evaluated. A pilot trial will assess the potential of this approach and provide information necessary to perform a cluster-randomized controlled trial (RCT). The cluster-randomized controlled trial (RCT) will together with qualitative interviews and observations, evaluate the effectiveness of the intervention. Outcomes will be measured at baseline (September /October 2016) at the end of the intervention which lasts for 7 months (May 2017), and 1 year after the end of the intervention (May 2018)

ELIGIBILITY:
Inclusion Criteria:

* Attends first grade in one of the ASPs included

Exclusion Criteria:

* Does not attend first grade in one of the ASPs included

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 456 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in minutes spent in moderate to vigorous physical activity in after school programs from baseline to end of intervention (7 months) and 1 year after end of intervention. | Baseline, end of intervention (7 months), 1 year after intervention
  Measures at baseline of a cluster randomized controlled intervention study and measures at the end of the 7 month intervention (measures of change) and 1 year after the end of the intervention (long-term effects). Physical activity is measured objectively by accelerometer (ActiGraph GM3X and GM3X+).

SECONDARY OUTCOMES:
Heath-related quality of life | Baseline, end of intervention (7 months), 1 year after intervention
  Parent-reported, measured by KIDSCREEN-27 questionnaire (parent version)
Leisure time physical activity | Baseline, end of intervention (7 months), 1 year after intervention
  Self-reported/parent-reported, measured by UngKan-2 questionnaire
Active play in the ASP | Baseline, end of intervention (7 months), 1 year after intervention
  Self-reported/parent-reported, measured by questionnaire
Body mass index | Baseline, end of intervention (7 months), 1 year after intervention
  kg/(m2), height and weight measured objectively
Physical activity and play (observations) | Baseline or end of intervention (7 months)
  Qualitative observations of physical activity and play among children during one day in the ASP (sub sample)
Physical activity and play (interviews) | End of intervention (7 months)
  Qualitative interviews with children about active play and physical activity in ASP (sub sample)

OTHER OUTCOMES:
Work-related Basic Need Satisfaction among SFP-staff | Baseline, end of intervention (7 months), 1 year after intervention
  Self-reported, measured by the Work-related Basic Need Satisfaction Scale (W-BNS)
Work motivation in ASP-staff | Baseline, end of intervention (7 months), 1 year after intervention
  Self-reported, measured by the Multidimensional Work Motivation Scale (MWMS)
Job Satisfaction in ASP-staff | Baseline, end of intervention (7 months), 1 year after intervention
  Self-reported, measured by the Job Satisfaction Scale (JSS)
Satisfaction with Life in ASP-staff | Baseline, end of intervention (7 months), 1 year after intervention
  Self-reported, measured by the Satisfaction with Life Scale (SWSL)
ASP-staff's experiences of taking part in the intervention (process outcome) | End of intervention (7 months)
  Focus group interviews (sub sample)
Local physiotherapist's experiences of taking part in the intervention (process outcome) | End of intervention (7 months)
  Focus group interviews

CONTACTS AND LOCATIONS:
Overall Officials: Kirsti Riiser, Phd, Principal Investigator — Oslo Metropolitan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riiser K, Richardsen KR, Haugen ALH, Lund S, Londal K. Active play in ASP -a matched-pair cluster-randomized trial investigating the effectiveness of an intervention in after-school programs for supporting children's physical activity. BMC Public Health. 2020 Apr 15;20(1):500. doi: 10.1186/s12889-020-08645-1. PMID 32295569
- [Derived] Riiser K, Helseth S, Ellingsen H, Fallang B, Londal K. Active Play in After-school Programmes: development of an intervention and description of a matched-pair cluster-randomised trial assessing physical activity play in after-school programmes. BMJ Open. 2017 Aug 4;7(8):e016585. doi: 10.1136/bmjopen-2017-016585. PMID 28780558